CLINICAL TRIAL: NCT00197470
Title: Effects of Pro-Inflammatory and Anti-Inflammatory Cytokine Gene Polymorphism on the Development of Gastric Cancer and Peptic Ulcer in Japanese
Brief Title: Cytokine Gene Polymorphisms in Gastric Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamamatsu University (Other)
Collaborators: Yokoyama Foundation for Clinical Pharmacology (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Mitsu-001
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Gastric Ulcer; Duodenal Ulcer; Gastric Cancer
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer; Stomach Neoplasms | interventions — Interleukin-1; Tumor Necrosis Factor-alpha; Interleukin-10

INTERVENTIONS:
Procedure: IL-1, TNF-alpha, Il-10

SUMMARY:
Recently, cytokine polymorphisms are considered to play an important role in the pathogenesis of peptic ulcer and gastric cancer. We intended to clarify the association between polymorphisms of pro-inflammatory and anti-inflammatory cytokines, and the susceptibility to gastric cancer, gastric ulcer and duodenal ulcer in Japan, and to detect the individuals who have higher risks for gastrointestinal disease development.

DETAILED DESCRIPTION:
H. pylori infection has close associations with the development of peptic ulcer diseases as well as gastric cancer, gastric adenoma, and gastric MALT lymphoma. The association of the host genetics with the susceptibility to various gastroduodenal disorders has been intensively investigated in the pathogenesis of peptic ulcer and gastric cancer by H. pylori infection .

In chronic active gastritis induced by H. pylori infection, activated neutrophils and mononuclear cells produce several pro-inflammatory and anti-inflammatory cytokines. In fact, levels of pro-inflammatory and anti-inflammatory cytokines are elevated in gastric mucosa infected with H. pylori.

Cytokine polymorphisms are associated with various inflammatory and autoimmune diseases. Recently, cytokine polymorphisms are considered to play an important role in the pathogenesis of peptic ulcer and gastric cancer. However, the roles of the IL-10 polymorphisms on the pathogenesis of H. pylori-related gastric cancer and peptic ulcer have not been fully elucidated.It is unclear whether pro-inflammatory and anti-inflammatory cytokines polymorphisms were associated with pathogenesis of peptic ulcer and gastric cancer in Japan. Then, we intended to clarify the association between polymorphisms of IL-10 and the susceptibility to gastric cancer, gastric ulcer and duodenal ulcer in Japan, and to detect the individuals who have higher risks for gastrointestinal disease development.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* patinets without H. pylori

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-01

CONTACTS AND LOCATIONS:
Overall Officials: MItsushige Sugimoto, Study Chair — First department of medicine, Hamamatsu University School of medicine
Locations (1):
- Hamamatsu University School of Medicine, Hamamatsu, Japan